CLINICAL TRIAL: NCT04415073
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Axatilimab for the Treatment of Hospitalized Patients With Respiratory Signs and Symptoms Secondary to Novel Coronavirus Disease (COVID-19)
Brief Title: A Phase 2 Study to Evaluate Axatilimab for Hospitalized Participants With Respiratory Involvement Secondary to COVID-19
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Given enrollment challenges, partly attributable to the constantly changing COVID-19 treatment landscape, the trial has been closed.
Sponsor: Syndax Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SNDX-6352-0505
Record Dates: First submitted 2020-05-29; First posted 2020-06-04 (Actual); Results first posted 2022-07-22 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-06

CONDITIONS: Coronavirus; COVID; ARDS; Cytokine Storm; Cytokine Release Syndrome
MeSH Terms: conditions — Coronavirus Infections; Cytokine Release Syndrome | interventions — axatilimab

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Axatilimab (SNDX-6352) (Active Comparator): Axatilimab on Days 1 and 15, IV + SOC
  Interventions: Drug: SNDX-6352
- Placebo (Placebo Comparator): Matching placebo on Days 1 and 15, IV + SOC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SNDX-6352 — SNDX-6352
  Other Names: Axatilimab
  Arms: Axatilimab (SNDX-6352)
Drug: Placebo — Placebo comparator
  Arms: Placebo

SUMMARY:
This was a randomized, double-blind, placebo-controlled, 29-day study to assess the efficacy and safety of axatilimab plus standard of care (SOC), compared with placebo plus SOC, in participants with respiratory signs and symptoms secondary to COVID-19.

DETAILED DESCRIPTION:
Axatilimab (SNDX-6352) is a humanized immunoglobin G4 monoclonal antibody with high affinity against colony stimulating factor-1 receptor (CSF-1R) under investigation for the prevention or treatment of respiratory signs and symptoms secondary to COVID-19.

This was a Phase 2, randomized, double-blind, placebo-controlled, multicenter study to evaluate the efficacy, safety and tolerability of axatilimab as an add-on to SOC therapy in hospitalized participants with respiratory signs and symptoms secondary to COVID-19 compared to SOC treatment.

Eligible participants were to be randomized in a 1:1 ratio to 1 of 2 treatment groups, active or control. All participants were to receive axatilimab or matching placebo intravenously (IV) as an add-on to SOC on Day 1, within 8 hours of randomization and on Day 15. Participants were to be followed for at least 28 days (+3 days) after the first dose of study intervention (Day 29).

The primary objective of the study was to assess the proportion of participants alive and free of respiratory failure at Day 29.

ELIGIBILITY:
Inclusion Criteria:

Type of Participant and Disease Characteristics -

1. Documented or confirmed severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection by an FDA-approved polymerase chain reaction test of nasopharyngeal swab or stool less than 72 hours before randomization
2. Hospitalized for COVID-19
3. Illness of any duration with at least 1 of the following:

   1. Clinical assessment (evidence of rales/crackles on exam) and peripheral capillary oxygen saturation less than or equal to 94% on room air, or
   2. Requiring mechanical ventilation and/or supplemental oxygen, or
   3. Radiographic evidence (chest x-ray or computed tomography scan) of 1 of the following:

      * Ground-glass opacities, or
      * Local or bilateral patchy infiltrates, or
      * Interstitial pulmonary infiltrates
4. If the participant was intubated, must have been intubated less than 24 hours prior to randomization

   Sex and Contraception Guidelines -
5. Contraceptive use by men or women should have been consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

   Informed Consent -
6. Capable of giving signed informed consent or by a designated representative, which includes compliance with the requirements and restrictions listed in the informed consent form and in this protocol

Exclusion Criteria:

Medical Conditions -

1. Active bacterial pneumonia defined: based on either lobar consolidation on x-ray, positive sputum cultures, or leukocytosis with a left shift
2. Known active tuberculosis
3. Participants with acquired immune deficiency syndrome
4. It is not in the best interest of the participants to participate, in the opinion of the treating Investigator.
5. In the opinion of the investigator, progression to death was imminent and inevitable within the next 24 hours, irrespective of the provision of treatments.
6. Female participants who were pregnant or breastfeeding or expecting to conceive within the projected duration of the study, starting with the screening visit through 90 days after the last dose of study intervention

   Excluded Prior/Concomitant Therapy -
7. Prior treatment with other agents with actual or possible direct acting anti-inflammatory activity against SARS-CoV-2 in the past 30 days (for example, chloroquine, hydroxychloroquine)
8. Treatment with convalescent plasma
9. Treatment with high doses of corticosteroids (greater than 20 milligrams daily, prednisone equivalent) prior to randomization
10. Treatment with immunomodulators including anti-interleukin (IL)-6, anti-IL-6 receptor antagonists, or with Janus kinase inhibitors in the past 30 days or plans to receive during the study period
11. Previous exposure to study intervention or any other agent targeting colony stimulating factor-1 or CSF-1R or known allergy/sensitivity to study intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-05-30 (Actual); Primary Completion 2020-07-13 (Actual); Study Completion 2020-07-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - HonorHealth, Scottsdale, Arizona
  - Montefiore Medical Center, The Bronx, New York

REFERENCES:
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was terminated by the Sponsor given enrollment challenges, partly attributable to the constantly changing novel coronavirus disease (COVID-19) treatment landscape. Due to study termination and only 1 participant being enrolled there are concerns regarding participant confidentiality, therefore no data are being reported.
Groups:
- Axatilimab (SNDX-6352): Axatilimab on Days 1 and 15, intravenous (IV) + standard of care (SOC)
Period: Overall Study
Arm/Group | Axatilimab (SNDX-6352) | Placebo
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This study was terminated by the Sponsor. Due to study termination and only 1 participant being enrolled there are concerns regarding participant confidentiality, therefore no data are being reported.
Groups:
- Total: Total of all reporting groups
Arm/Group | Axatilimab (SNDX-6352) | Placebo | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Continuous
Sex: Female, Male
Ethnicity (NIH/OMB)
Race (NIH/OMB)
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Count Of Participants Alive And Free Of Respiratory Failure At Day 29
Description: Respiratory failure was defined by need for mechanical ventilation, extracorporeal membrane oxygenation, non-invasive ventilation >6 liters oxygen/minute, or clinical diagnosis of respiratory failure with initiation of none of these measures only when clinical decision-making was driven solely by resource limitation.
Time Frame: Day 29
Population: as for baseline characteristics
Arm/Group | Axatilimab (SNDX-6352) | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Count Of Participants With Secondary Clinical Improvement Outcomes At Day 29
Description: Participants achieving a ≥2 category improvement on a 7-point ordinal score relative to the baseline on Day 28 as collected on Day 29 are reported.
Time Frame: Day 29
Population: as for baseline characteristics
Arm/Group | Axatilimab (SNDX-6352) | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Time To Clinical Improvement
Description: The time to clinical improvement is defined as a national early warning score of ≤2 maintained for 24 hours.
Time Frame: Baseline through Day29
Population: as for baseline characteristics
Arm/Group | Axatilimab (SNDX-6352) | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change From Baseline At Day 29 In Oxygenation In Hospitalized Adults With Respiratory Signs And Symptoms Secondary To COVID-19 Treated With Axatilimab
Description: The change from baseline at Day 29 or hospital discharge or death, if sooner, in the ratio of peripheral hemoglobin oxygen saturation to fraction of inspired oxygen is evaluated.
Time Frame: Baseline, Day 29
Population: as for baseline characteristics
Arm/Group | Axatilimab (SNDX-6352) | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change From Baseline At Day 15 In Biomarkers Following Treatment With Axatilimab
Description: The change from baseline at Day 15 in serum concentrations of interleukin 6 and c-reactive protein or hospital discharge or death is evaluated.
Time Frame: Baseline, Day 15
Population: as for baseline characteristics
Arm/Group | Axatilimab (SNDX-6352) | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Count Of Participants Experiencing Adverse Events And Serious Adverse Events
Description: This outcome measure evaluates the safety and tolerability of axatilimab within the same population. A summary of all serious adverse events and other adverse events (nonserious) regardless of causality is located in the 'Reported Adverse Events' section.
Time Frame: Baseline through Day 29
Population: as for baseline characteristics
Arm/Group | Axatilimab (SNDX-6352) | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Count Of Participants Requiring Ventilation Support
Description: Participants who required initiation of mechanical ventilation after study entry are analyzed.
Time Frame: Baseline through Day 29
Population: as for baseline characteristics
Arm/Group | Axatilimab (SNDX-6352) | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Count Of Participants Considered Severe Acute Respiratory Syndrome Coronavirus (SARS-CoV-2) Free By Day 15
Description: This outcome measure evaluates the antiviral effects of axatilimab in hospitalized adults by Day 15 or hospital discharge, whichever was sooner, with recently diagnosed SARS-CoV-2 infection.
Time Frame: Day 15
Population: as for baseline characteristics
Arm/Group | Axatilimab (SNDX-6352) | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Pharmacokinetics: Serum Concentration Of Axatilimab And Anti-drug Antibodies
Description: The serum concentration of axatilimab and presence of anti-drug antibodies is evaluated.
Time Frame: Day 29
Population: as for baseline characteristics
Arm/Group | Axatilimab (SNDX-6352) | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: This study was terminated by the Sponsor. Due to study termination and only 1 participant being enrolled there are concerns regarding participant confidentiality, therefore no data are being reported.
Description: This study was terminated by the Sponsor. Due to study termination and only 1 participant being enrolled there are concerns regarding participant confidentiality, therefore no data are being reported.
Arm/Group | Axatilimab (SNDX-6352) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This study was terminated by the Sponsor given enrollment challenges, partly attributable to the constantly changing COVID-19 treatment landscape. Due to study termination and only 1 participant being enrolled there are concerns regarding participant confidentiality, therefore no data are being reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-23): https://cdn.clinicaltrials.gov/large-docs/73/NCT04415073/Prot_SAP_000.pdf